CLINICAL TRIAL: NCT00940719
Title: The Effects of Vitamin D3 Supplementation on the T Cell Compartment in Multiple Sclerosis; a Pilot Study
Brief Title: Vitamin D3 Supplementation and the T Cell Compartment in Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Orbis Medical Centre (Other)
Responsible Party: Prof. dr. Raymond Hupperts, M.D., Ph.D., Orbis Medical Center Sittard, Maastricht University Medical Center Maastricht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MUMC09T43
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Regulatory T cell function; Vitamin D; Vitamin D3; 25-hydroxyvitamin D
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D3 (Experimental): Patients receive 1dd 500ug vitamin D3 for 3 months
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D3 — Oil-based solution, 1 dose of 500 microgram each day, during 3 months.
  Other Names: Vigantol Oil (Merck)

SUMMARY:
In patients with Relapsing Remitting Multiple Sclerosis (RRMS), the investigators observed a positive correlation between regulatory T cell (Treg) function and vitamin D status. The present goal is to assess whether Treg function improves on supplementation with vitamin D3.

DETAILED DESCRIPTION:
In several studies, Multiple Sclerosis (MS) incidence and disease activity has been related with vitamin D status. We observed that RRMS patients who remained relapse free before blood collection had a better vitamin D status than patients who experienced relapses (Smolders et al. Mult Scler 2008;17:1220-1224). Since vitamin D3 is a potent promotor of T cell regulation in vitro (Smolders et al. J Neuroimmunol 2008;194:7-17), we hypothesised that a promotion of Treg function in MS patients might underlie its association with MS disease activity. In a cohort of RRMS patients, we observed a positive correlation of Treg function with vitamin D status (Smolders et al. PLoS ONE 2009;4:e6635). Furthermore, vitamin D status correlated positively with a Th1/Th2-balance which was more directed towards Th2. In the present study, we will assess whether treatment of RRMS patients with vitamin D3 promotes T cell regulation.

In the present study, RRMS patients will be supplemented with vitamin D3, and regulatory T cell tests will be performed before and after supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing Remitting MS (Revised MCDonald criteria 2005)
* Age > 18 years

Exclusion Criteria:

* Progressive MS phenotype
* Abnormalities of vitamin D hormonal system other than low dietary intake or limited sun exposure
* Intake of drugs that influence vitamin D homeostasis other than corticosteroids
* Conditions with in increased susceptibility to hypercalcemia
* Alcohol or drug abuse
* Pregnancy or the intention to become pregnant within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
T cell regulation | 3 months

SECONDARY OUTCOMES:
serum 25-hydroxyvitamin D levels | 3 months
calcium metabolism | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Hupperts, M.D., Ph.D., Study Director — Orbis Medical Center Sittard, Maastricht Univeristy Medical Center Maastricht; Joost Smolders, M.D., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Orbis Medical Center, Sittard, Netherlands

REFERENCES:
- [Background] Smolders J, Menheere P, Kessels A, Damoiseaux J, Hupperts R. Association of vitamin D metabolite levels with relapse rate and disability in multiple sclerosis. Mult Scler. 2008 Nov;14(9):1220-4. doi: 10.1177/1352458508094399. Epub 2008 Jul 24. PMID 18653736
- [Background] Smolders J, Damoiseaux J, Menheere P, Hupperts R. Vitamin D as an immune modulator in multiple sclerosis, a review. J Neuroimmunol. 2008 Feb;194(1-2):7-17. doi: 10.1016/j.jneuroim.2007.11.014. Epub 2008 Jan 4. PMID 18177949
- [Background] Smolders J, Thewissen M, Peelen E, Menheere P, Tervaert JW, Damoiseaux J, Hupperts R. Vitamin D status is positively correlated with regulatory T cell function in patients with multiple sclerosis. PLoS One. 2009 Aug 13;4(8):e6635. doi: 10.1371/journal.pone.0006635. PMID 19675671
- [Background] Smolders J, Menheere P, Thewissen M, Peelen E, Tervaert JW, Hupperts R, Damoiseaux J. Regulatory T cell function correlates with serum 25-hydroxyvitamin D, but not with 1,25-dihydroxyvitamin D, parathyroid hormone and calcium levels in patients with relapsing remitting multiple sclerosis. J Steroid Biochem Mol Biol. 2010 Jul;121(1-2):243-6. doi: 10.1016/j.jsbmb.2010.03.001. Epub 2010 Mar 6. PMID 20211254
- [Derived] Smolders J, Peelen E, Thewissen M, Cohen Tervaert JW, Menheere P, Hupperts R, Damoiseaux J. Safety and T cell modulating effects of high dose vitamin D3 supplementation in multiple sclerosis. PLoS One. 2010 Dec 13;5(12):e15235. doi: 10.1371/journal.pone.0015235. PMID 21179201